CLINICAL TRIAL: NCT03045432
Title: Passive Range of Motion and Position Training for Stroke Patients With Hemiplegia to Prevent Shoulder Injury or Pain- Ultrasonographic Study
Brief Title: Shoulder Passive Range of Motion and Positioning Exercise on Hemiplegic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMRPG866091
Record Dates: First submitted 2017-02-05; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Shoulder Pain; Hemiplegia; Stroke; Rotator Cuff Injury
Keywords: Stroke; Hemiplegia; Rotator Cuff Injury
MeSH Terms: conditions — Shoulder Pain; Hemiplegia; Stroke; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video-teaching materials (Experimental): * regular passive ROM exercise
  * regular rehabilitation programe
  * alternative video-teaching materials
  Interventions: Other: video-teaching; Other: oral-teaching; Other: regular rehabilitation program
- control group (Other): * regular passive ROM exercise
  * regular rehabilitation programe
  * regular oral-teaching materials
  Interventions: Other: oral-teaching; Other: regular rehabilitation program

INTERVENTIONS:
Other: video-teaching — By watching a video specially designed by a rehabilitation team, the participants may learn how to position their affected arm properly (30 minutes per time, twice a day for five days in a week), how to transfer safely with the help from the caregivers, how to execute appropriate passive range of motion exercises regularly (15 minutes per time, twice a day for five days in a week), and be taught to be aware of not doing insecure pulley exercises nor carrying stuffs which are too heavy.
  Arms: video-teaching materials
Other: oral-teaching — The nurses will teach patients how to position their affected arm properly, how to transfer safely with the help from the caregivers, how to execute appropriate passive range of motion exercises regularly, and be taught to be aware of not doing insecure pulley exercises nor carrying stuffs which are too heavy on the admission date of hospitalization.
Other: regular rehabilitation program — Regular occupational therapy program and regular physical therapy program in the rehabilitation department of the hospital.

SUMMARY:
Several factors associated with the hemiplegic shoulder pain after stroke includes rotator cuff injury, bicipital tendonitis, impingement, spasticity, limited external rotation of shoulder joint, adhesive capsulitis, shoulder subluxation, shoulder hand syndrome, and brachial/axillary neuropathy. In this study, the investigators aim to usie high frequency ultrasound to evaluate the relationship between stroke patients with poor shoulder motor function and shoulder tendon injury. Also, assumed that performing passive range of motion and positioning training might prevent tendon injury of shoulder and hemiplegic shoulder pain in either acute or chronic stage of stroke.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is a common complication. Several factors associated with the hemiplegic shoulder pain includes rotator cuff injury, bicipital tendonitis, impingement, spasticity, limited external rotation of shoulder joint, adhesive capsulitis, shoulder subluxation, shoulder hand syndrome, and brachial/axillary neuropathy. Flaccidity has a positive association with soft tissue injury or tendon injury of the shoulder.

In the preliminary study, base on the sonography results, it is found that the possibility of getting tendon injury or inflammation on the affected shoulder joint is higher in the group of patients who were with worse motor functions during the rehabilitation in hospital.

In this study, one hundred acute stroke patients with hemipelgia will be enrolled. And those participants would be separated into 2 groups: control group (Brunnstrom stage IV-VI) and experimental group (Brunnstrom stage I-III). Clinical characteristics and physical findings will be recorded on the admission date. During the process, the investigators will use high frequency (5-12 MHz) musculoskeletal ultrasound to evaluate those tendons around bilateral shoulder joints on the admission date and at 2 weeks later. In the first year after stroke, half patients in those 2 groups will perform positioning training and passive range of motion for affected shoulder either during hospitalization or after being discharged. Then, the investigators will execute physical examination and use high frequency ultrasound to evaluate those tendons around bilateral shoulder joints of the participants twice after 6 months and 12 months. Then, the investigators will discuss the incidences of shoulder tendon injury after receiving rehabilitation program according to ultra-sonographic findings.

ELIGIBILITY:
Inclusion Criteria:

* stroke with hemiplegia
* age between 18-80

Exclusion Criteria:

* recurrent stoke patient
* previous history of shoulder pain, any injuries and operation in shoulder joint, frozen shoulder, tendinitis in shoulder joint,
* any other systemic neuromuscular disease
* cognition or language impairment leading to communication difficulty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2009-06-30 (Actual)

PRIMARY OUTCOMES:
the change from baseline on hemiplegic upper extremity sonography | baseline (before intervention), changes from baseline sonography results at one week before being discharged and at six month after.
  A doctor will use a high frequency(5-12 MHz) sonography examination machine(Terason t300, Teratech Co., USA) as the evaluation tool of this study. The target muscles and structures around affected shoulder includes biceps, supraspinatus, infraspinatus, subscapularis, sub-deltoid bursa and ACJ.

SECONDARY OUTCOMES:
Brunnstrom motor recovery stage for motor ability | baseline (before intervention), changes from baseline Brunnstrom stage at one week before being discharged and at six month after.
  A physical therapist will measure Brunnstrom motor recovery stage and see the improvement of it from baseline till one week before being discharged and after six months.
Modified Ashworth scale for level of spasticity of affected arm | baseline (before intervention), changes from baseline level of spasticity at one week before being discharged and at six month after.
  A physical therapist will measure the level of spasticity in affected arm by using modified Ashworth scale.
Range of motion | baseline (before intervention), changes from baseline range of motions at one week before being discharged and at six month after.
  A physical therapist will measure range of motions of affected arm by using goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chi Huang, Bachelor, Principal Investigator — Study Principal Investigator ChangGungMH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Najenson T, Yacubovich E, Pikielni SS. Rotator cuff injury in shoulder joints of hemiplegic patients. Scand J Rehabil Med. 1971;3(3):131-7. No abstract available. PMID 5156175
- [Background] Griffin JW. Hemiplegic shoulder pain. Phys Ther. 1986 Dec;66(12):1884-93. doi: 10.1093/ptj/66.12.1884. PMID 2431421
- [Background] Bohannon RW, Larkin PA, Smith MB, Horton MG. Shoulder pain in hemiplegia: statistical relationship with five variables. Arch Phys Med Rehabil. 1986 Aug;67(8):514-6. PMID 3741075
- [Background] Turner-Stokes L, Jackson D. Shoulder pain after stroke: a review of the evidence base to inform the development of an integrated care pathway. Clin Rehabil. 2002 May;16(3):276-98. doi: 10.1191/0269215502cr491oa. PMID 12017515
- [Background] Snels IA, Dekker JH, van der Lee JH, Lankhorst GJ, Beckerman H, Bouter LM. Treating patients with hemiplegic shoulder pain. Am J Phys Med Rehabil. 2002 Feb;81(2):150-60. doi: 10.1097/00002060-200202000-00013. PMID 11807352
- [Background] Van Ouwenaller C, Laplace PM, Chantraine A. Painful shoulder in hemiplegia. Arch Phys Med Rehabil. 1986 Jan;67(1):23-6. PMID 3942479
- [Background] Gilmore PE, Spaulding SJ, Vandervoort AA. Hemiplegic shoulder pain: implications for occupational therapy treatment. Can J Occup Ther. 2004 Feb;71(1):36-46. doi: 10.1177/000841740407100108. PMID 15015899
- [Background] Snels IA, Beckerman H, Twisk JW, Dekker JH, Peter De Koning, Koppe PA, Lankhorst GJ, Bouter LM. Effect of triamcinolone acetonide injections on hemiplegic shoulder pain : A randomized clinical trial. Stroke. 2000 Oct;31(10):2396-401. doi: 10.1161/01.str.31.10.2396. PMID 11022070
- [Background] Parker VM, Wade DT, Langton Hewer R. Loss of arm function after stroke: measurement, frequency, and recovery. Int Rehabil Med. 1986;8(2):69-73. doi: 10.3109/03790798609166178. PMID 3804600
- [Background] Wanklyn P, Forster A, Young J. Hemiplegic shoulder pain (HSP): natural history and investigation of associated features. Disabil Rehabil. 1996 Oct;18(10):497-501. doi: 10.3109/09638289609166035. PMID 8902421
- [Background] Lo SF, Chen SY, Lin HC, Jim YF, Meng NH, Kao MJ. Arthrographic and clinical findings in patients with hemiplegic shoulder pain. Arch Phys Med Rehabil. 2003 Dec;84(12):1786-91. doi: 10.1016/s0003-9993(03)00408-8. PMID 14669184
- [Background] Ikai T, Tei K, Yoshida K, Miyano S, Yonemoto K. Evaluation and treatment of shoulder subluxation in hemiplegia: relationship between subluxation and pain. Am J Phys Med Rehabil. 1998 Sep-Oct;77(5):421-6. doi: 10.1097/00002060-199809000-00012. PMID 9798835
- [Background] Poulin de Courval L, Barsauskas A, Berenbaum B, Dehaut F, Dussault R, Fontaine FS, Labrecque R, Leclerc C, Giroux F. Painful shoulder in the hemiplegic and unilateral neglect. Arch Phys Med Rehabil. 1990 Aug;71(9):673-6. PMID 2375673
- [Background] Ada L, Goddard E, McCully J, Stavrinos T, Bampton J. Thirty minutes of positioning reduces the development of shoulder external rotation contracture after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2005 Feb;86(2):230-4. doi: 10.1016/j.apmr.2004.02.031. PMID 15706548
- [Background] Ada L, Foongchomcheay A, Canning C. Supportive devices for preventing and treating subluxation of the shoulder after stroke. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003863. doi: 10.1002/14651858.CD003863.pub2. PMID 15674917
- [Background] Chae J, Mascarenhas D, Yu DT, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Fang ZP. Poststroke shoulder pain: its relationship to motor impairment, activity limitation, and quality of life. Arch Phys Med Rehabil. 2007 Mar;88(3):298-301. doi: 10.1016/j.apmr.2006.12.007. PMID 17321820
- [Background] Dekker JH, Wagenaar RC, Lankhorst GJ, de Jong BA. The painful hemiplegic shoulder: effects of intra-articular triamcinolone acetonide. Am J Phys Med Rehabil. 1997 Jan-Feb;76(1):43-8. doi: 10.1097/00002060-199701000-00008. PMID 9036910
- [Background] Lindgren I, Jonsson AC, Norrving B, Lindgren A. Shoulder pain after stroke: a prospective population-based study. Stroke. 2007 Feb;38(2):343-8. doi: 10.1161/01.STR.0000254598.16739.4e. Epub 2006 Dec 21. PMID 17185637
- [Background] Brandt TD, Cardone BW, Grant TH, Post M, Weiss CA. Rotator cuff sonography: a reassessment. Radiology. 1989 Nov;173(2):323-7. doi: 10.1148/radiology.173.2.2678248.
- [Background] Crass JR, Craig EV, Feinberg SB. Ultrasonography of rotator cuff tears: a review of 500 diagnostic studies. J Clin Ultrasound. 1988 Jun;16(5):313-27. doi: 10.1002/jcu.1870160506. PMID 3152389
- [Background] van Holsbeeck MT, Kolowich PA, Eyler WR, Craig JG, Shirazi KK, Habra GK, Vanderschueren GM, Bouffard JA. US depiction of partial-thickness tear of the rotator cuff. Radiology. 1995 Nov;197(2):443-6. doi: 10.1148/radiology.197.2.7480690.
- [Background] Aras MD, Gokkaya NK, Comert D, Kaya A, Cakci A. Shoulder pain in hemiplegia: results from a national rehabilitation hospital in Turkey. Am J Phys Med Rehabil. 2004 Sep;83(9):713-9. doi: 10.1097/01.phm.0000138739.18844.88. PMID 15314536
- [Background] Lee CL, Chen TW, Weng MC, Wang YL, Cheng HS, Huang MH. Ultrasonographic findings in hemiplegic shoulders of stroke patients. Kaohsiung J Med Sci. 2002 Feb;18(2):70-6. PMID 12056171
- [Background] Pong YP, Wang LY, Wang L, Leong CP, Huang YC, Chen YK. Sonography of the shoulder in hemiplegic patients undergoing rehabilitation after a recent stroke. J Clin Ultrasound. 2009 May;37(4):199-205. doi: 10.1002/jcu.20573. PMID 19253350